CLINICAL TRIAL: NCT03363737
Title: Can Facebook Reduce Perceived Anxiety Among College Students? A Randomized Controlled Exercise Trial Using the Transtheoretical Model of Behavior Change
Brief Title: Transtheoretical Model of Behavior Change and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi, Oxford (Other)
Responsible Party: Principal Investigator, Paul D. Loprinzi, Associate Professor of Health and Exercise Science, University of Mississippi, Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-018
Record Dates: First submitted 2017-11-29; First posted 2017-12-06 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Psychological; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Transtheoretical Model

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static (Active Comparator)
  Interventions: Behavioral: Transtheoretical Model
- Dynamic (Experimental)
  Interventions: Behavioral: Transtheoretical Model

INTERVENTIONS:
Behavioral: Transtheoretical Model — Exposure to content on Facebook, either daily (dynamic) or just at one time period (static).

SUMMARY:
Examine the utility of the Transtheoretical Model in influencing anxiety among college students. Employ a randomized controlled intervention including a static and dynamic Facebook intervention. The static group accessed a Facebook page featuring 96 statuses. Statuses were intended to engage cognitive processes, followed by behavioral processes of change per the Transtheoretical Model of behavior change. Content posted on the static Facebook page was identical to the dynamic page. However, the static group viewed all 96 statuses on the first day of the study, while the dynamic group received only 1-2 of these status updates per day throughout the intervention. Anxiety was measured using the Overall Anxiety Severity and Impairment Scale (OASIS). Time spent engaging in physical activity was assessed using the International Physical Activity Questionnaire (IPAQ).

ELIGIBILITY:
Inclusion Criteria:

* Having an active Facebook account
* Daily access to a Smart Phone
* Current University of Mississippi email account

Exclusion Criteria:

* Outside the age range of 18-35

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Changes in Anxiety | At baseline and at the end of the 8-week intervention
  OASIS, Overall Anxiety Severity and Impairment Scale. There are 5 questions in this scale, with each question including 5 response options (ranging from 0-4). The total score is reported, which ranges from 0-20 (higher score indicates greater anxiety).

REFERENCES:
- [Derived] Frith E, Loprinzi P. Can Facebook Reduce Perceived Anxiety Among College Students? Randomized Controlled Exercise Trial Using the Transtheoretical Model of Behavior Change. JMIR Ment Health. 2017 Dec 8;4(4):e50. doi: 10.2196/mental.8086. PMID 29222077